CLINICAL TRIAL: NCT04013230
Title: Group Sessions and Web-based Treatment Targeting Children With Obesity Age 5-12 Years and Their Families - a Randomized Controlled Trial of Children With Obesity in Northern Sweden
Brief Title: Group Sessions and Web-based Treatment Targeting Children With Obesity Age 5-12 Years and Their Families
Acronym: Webcop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Västernorrland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02343
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; BMI SDS
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care according to regular treatment routines at the clinic.
  Interventions: Behavioral: Usual care; Behavioral: Web-COP
- Web-COP (Active Comparator): Usual care plus group sessions and a web-based treatment program
  Interventions: Behavioral: Usual care; Behavioral: Web-COP

INTERVENTIONS:
Behavioral: Usual care — Visit doctor and nurse at the clinic.
Behavioral: Web-COP — Usual care plus group sessions and a web-based treatment program for 12 weeks for the child and parents.

SUMMARY:
The aim of this study is to assess the efficacy of group sessions and a web-based program for children with obesity age 5-12 years and their parents.

The intervention consist of a doctor's appointment, four group-based education sessions over four weeks, psychical activity on prescription and a 12-week web-based treatment program and will be offered to children aged 5-12 years with obesity (International Obesity Task Force-BMI >30), and their parents.

DETAILED DESCRIPTION:
Obesity in children and adolescents worldwide has increased from 1 % in 1975 to about 6 % in 2016. Experts have estimated that the world will have more obese children and adolescents than underweight at the year 2022. Preventing and reversing excess weight gain in children is important since obesity often tracks into adulthood with adverse health consequences.

Web-based interventions have been shown to be effective, to have a beneficial treatment outcome and have been proposed to have great potential to reach many children and improve cost effectiveness.

This is a randomized controlled study with cross-over design. The intervention consist of a doctor's appointment, four group-based education sessions over four weeks, psychical activity on prescription and a 12-week web-based treatment program. The control group will have standard care treatment consisting of doctor's appointment and, in some cases, contact with dietician.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to International Obesity Task Force (IOTF)
* Be able to speak and write Swedish
* Have internet access in parents' home

Exclusion Criteria:

* Obesity together with other severe disease including neuropsychiatric disorder

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-08-21 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMI-SDS | At baseline, 2, 4 and 6 months
  Controll vs intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Arne Silfverdal, PhD, Principal Investigator — Umeå University
Locations (3):
- Sweden (3):
  - Outpatient peadictric clinic in Sollefteå hospital, Sollefteå
  - Outpatient peadiatric clinic in Sundsvalls hospital, Sundsvall
  - Umeå university, Umeå